CLINICAL TRIAL: NCT00193180
Title: Phase II Trial of Docetaxel Plus Imatinib Mesylate in Metastatic Breast Cancer
Brief Title: Docetaxel Plus Imatinib Mesylate in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 74
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Imatinib Mesylate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All patients in this study received docetaxel 30 mg/m2 weekly for 3 consecutive weeks of each 28-day cycle, along with continuous imatinib mesylate. Initially, imatinib mesylate was given at a dose of 600 mg orally daily, beginning concurrently with the first dose of docetaxel; however, after the first 15 patients were treated it became evident that this imatinib dose was not tolerable, and subsequent patients received imatinib mesylate 400 mg orally daily.
  Interventions: Drug: Imatinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Imatinib — Imatinib
  Other Names: Gleevec
Drug: Docetaxel — Docetaxel
  Other Names: Taxotere

SUMMARY:
This trial evaluates the novel combination of docetaxel with imatinib as first or second line therapy in advanced breast cancer with the aim of achieving higher effectiveness and potentially reducing side effects.

DETAILED DESCRIPTION:
All patients in this study received docetaxel 30 mg/m2 weekly for 3 consecutive weeks of each 28-day cycle, along with continuous imatinib mesylate. Initially, imatinib mesylate was given at a dose of 600 mg orally daily, beginning concurrently with the first dose of docetaxel; however, after the first 15 patients were treated it became evident that this imatinib dose was not tolerable, and subsequent patients received imatinib mesylate 400 mg orally daily

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Metastatic breast cancer confirmed by biopsy
* No more than one prior chemotherapy regimen for metastatic breast cancer
* Able to perform activities of daily living with minimal assistance
* Adequate bone marrow, liver and kidney function
* Age 18 years or older
* Give written informed consent

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Moderate to severe peripheral neuropathy
* Uncontrolled blood pressure or uncontrolled heart beat irregularities
* Diabetes Mellitus with fasting blood sugar greater than 200 mg %
* Significant heart disease within the prior 6 months
* Severe or uncontrolled medical disease
* Active uncontrolled infection
* Known chronic liver disease
* Known diagnosis of HIV infection
* Pregnant or breast feeding females

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-05; Primary Completion 2008-05 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - Tennessee Oncology, Nashville, Tennessee

REFERENCES:
- [Result] Yardley DA, Burris HA 3rd, Markus T, Spigel DR, Greco FA, Mainwaring M, Waterhouse DM, Webb CD, Hainsworth JD. Phase II trial of docetaxal plus imatinib mesylate in the treatment of patients with metastatic breast cancer. Clin Breast Cancer. 2009 Nov;9(4):237-42. doi: 10.3816/CBC.2009.n.040. PMID 19933079
- See also: Published article in Clinical Breast Cancer — http://cigjournals.metapress.com/content/hqr3590152282262/fulltext.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: All patients in this study received docetaxel 30 mg/m^2 weekly for 3 consecutive weeks of each 28-day cycle, along with continuous imatinib mesylate. Initially, imatinib mesylate was given at a dose of 600 mg orally daily, beginning concurrently with the first dose of docetaxel; however, after the first 15 patients were treated it became evident that this imatinib dose was not tolerable, and subsequent patients received imatinib mesylate 400 mg orally daily.
Period: Overall Study
Arm/Group | Intervention
Started | 37
Completed | 27
Not Completed | 10
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 8
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 59 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Defined as the proportion of patients with confirmed complete or partial response (CR or PR), recorded from date of treatment until date of recurrence or progressive disease, and assessed by RECIST v 1.1.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 37
percentage of participants | 16 [4.3 to 28.1]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the length of time, in months, that patients were alive from date of first protocol treatment until worsening of disease, assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intervention
Number analyzed (Participants) | 37
Months | 9.3 [3.7 to 13.6]

3. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from first protocol treatment to date of death due to any cause.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intervention
Number analyzed (Participants) | 37
months | 15.4 [9.6 to 26.7]

ADVERSE EVENTS:
Groups:
- Docetaxel+Imatinib: Patients received docetaxel 30mg/m2 IV weekly on days 1, 8, and 15 of each 28 day cycle. Patients received oral imatinib 400mg daily. Fifteen patients initially received oral imatinib 600mg daily but had their dose reduced to 400mg daily when they were unable to tolerate the higher dose.
Arm/Group | Docetaxel+Imatinib
Serious Adverse Events (participants affected / at risk) | 18/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel+Imatinib (N=37)
Infection - carcinomatous meningitis (Infections and infestations) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Rigors/chills (General disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (diverticular abscess) (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection - pneumonia (Infections and infestations) | 1 (5)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 1 (1)
Pain - abdomen (General disorders) | 1 (1)
Pain - chest (General disorders) | 1 (1)
Pain - pleura (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Renal failure (Renal and urinary disorders) | 1 (1)
Cardiac ischemia/infarction - rheumatic heart failure (Cardiac disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Thrombosis/embolism (vascular access) (Vascular disorders) | 1 (1) — Deep vein thrombosis
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel+Imatinib (N=37)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
ALT, SGPT (Metabolism and nutrition disorders) | 2 (7)
Altered mental status (Psychiatric disorders) | 2 (2)
AST, SGOT (Metabolism and nutrition disorders) | 2 (4)
Disease progression (carcinomatous meningitis) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Chills (Nervous system disorders) | 5 (7)
Confusion (Nervous system disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Dehydration (Gastrointestinal disorders) | 7 (7)
Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Dizziness (Nervous system disorders) | 3 (7)
Dysgeusia (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (27)
Edema - periorbital (Blood and lymphatic system disorders) | 2 (3)
Fever (General disorders) | 6 (8)
Hot flashes (Endocrine disorders) | 6 (32)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (42)
Hyperlacrimation (Eye disorders) | 7 (19)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 8 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Infection - herpes zoster (Infections and infestations) | 2 (2)
Infection - pneumonia (Infections and infestations) | 3 (5)
Infection - thrush (Infections and infestations) | 3 (5)
Infection - urinary tract (Infections and infestations) | 2 (2)
Insomnia (General disorders) | 4 (8)
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 (8)
Leukocytes (Blood and lymphatic system disorders) | 14 (42)
Lymphedema (Blood and lymphatic system disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 14 (19)
Myalgia (General disorders) | 10 (29)
Nail changes (Skin and subcutaneous tissue disorders) | 4 (10)
Neuropathy (Nervous system disorders) | 10 (32)
Night sweats (General disorders) | 2 (7)
Pain - abdomen (General disorders) | 4 (4)
Pain - chest (General disorders) | 3 (7)
Pain - headache (General disorders) | 4 (5)
Pain - joint (General disorders) | 2 (2)
Pain - limb (General disorders) | 2 (2)
Pain - throat (General disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Gastroesophageal reflux disorder (Gastrointestinal disorders) | 3 (3)
Taste alteration (Gastrointestinal disorders) | 6 (18)
Thrombus/thrombosis/embolism (Vascular disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Weakness (General disorders) | 6 (15)
Alopecia (General disorders) | 11 (50)
Hemoglobin (Blood and lymphatic system disorders) | 31 (113)
Anorexia (Gastrointestinal disorders) | 19 (52)
Constipation (Gastrointestinal disorders) | 15 (44)
Diarrhea (Gastrointestinal disorders) | 26 (71)
Fatigue (General disorders) | 31 (112)
Allergic reaction (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 30 (90)
Neutrophils (Blood and lymphatic system disorders) | 11 (22)
Pain - NOS (General disorders) | 17 (60)
Neuropathy - sensory (Nervous system disorders) | 8 (28)
Platelets (Blood and lymphatic system disorders) | 10 (12)
Vomiting (Gastrointestinal disorders) | 22 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.